CLINICAL TRIAL: NCT03637517
Title: Relative Bioavailability and Effect of Food on DSM265-TPGS 34% SDD Powder in Healthy Adult Subjects
Brief Title: Malaria: Relative Bioavailability and Food Effect of DSM265
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MMV_DSM265_18_01; B19-227 (Other: AbbVie)
Record Dates: First submitted 2018-08-15; First posted 2018-08-20 (Actual); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — DSM265

STUDY DESIGN:
Intervention Model Description: Phase 1, single-dose, open-label, randomized, parallel group design in healthy adults (males, females of non child bearing potential) in 3 groups of 14 subjects each.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DSM265-TPGS 34% SDD, 400 mg fasted (Experimental): Spray dried dispersion (SDD) formulation, powder containing 34.25% DSM265-TPGS (tocopheryl polyethylene glycol succinate)
  Interventions: Drug: DSM265-TPGS 34% SDD, 400 mg fasted
- DSM265-TPGS 34% SDD, 400 mg fed (Active Comparator): Spray dried dispersion (SDD) formulation, powder containing 34.25% DSM265-TPGS (tocopheryl polyethylene glycol succinate)
  Interventions: Drug: DSM265-TPGS 34% SDD, 400 mg fed
- DSM265 25% SDD, 400 mg fasted (Active Comparator): Spray dried dispersion (SDD) formulation, powder containing 25% DSM265 as free base
  Interventions: Drug: DSM265 25% SDD, 400 mg fasted

INTERVENTIONS:
Drug: DSM265-TPGS 34% SDD, 400 mg fasted — New formulation allowing smaller volumes of dissolution in a common vehicle (water), administered to subjects in a fasted state.
  Other Names: DSM265
  Arms: DSM265-TPGS 34% SDD, 400 mg fasted
Drug: DSM265-TPGS 34% SDD, 400 mg fed — New formulation allowing smaller volumes of dissolution in a common vehicle (water), administered to subjects in a fed state.
  Other Names: DSM265
  Arms: DSM265-TPGS 34% SDD, 400 mg fed
Drug: DSM265 25% SDD, 400 mg fasted — Reference formulation used in early clinical trials.
  Other Names: DSM265
  Arms: DSM265 25% SDD, 400 mg fasted

SUMMARY:
Phase 1 study designed to evaluate the relative bioavailability of a single dose of a test formulation, DSM265-TPGS 34% SDD powder in comparison with a reference DSM265 25% SDD powder formulation used in early clinical trials.

DETAILED DESCRIPTION:
The objective of this study is to compare the relative bioavailability of oral DSM265-TPGS 34% SDD formulation with that of a reference 25% SDD powder for suspension used in previous clinical trials. Another objective of the study is to evaluate the effect of food on bioavailability of the DSM265-TPGS 34% SDD formulation.

The current 25% SDD powder for suspension clinical formulation is a suspension which requires reconstitution/administration in 240 mL sucralose based vehicle (for a 400 mg adult dose). This volume is too large for paediatric patients with malaria (e.g., translates into a 30 mL volume for 0.5-2 yr old patients); also, the dosing vehicle is not commercially viable. The new formulation dissolves in a smaller volume of a more common vehicle, water (40 mL for 400 mg adult dose).

ELIGIBILITY:
1. Subjects or their legally authorized representative must voluntarily sign and date each informed consent, approved by an Independent Ethics Committee(IEC) / Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.
2. Male or female between 18 and 55 years of age inclusive at the time of screening.
3. Body Mass Index (BMI) is ≥ 18.0 to ≤ 29.9 kg/m2 after rounding to the tenths decimal. BMI is calculated as weight in kg divided by the square of height measured in meters.
4. Females must be of Non-Childbearing Potential as defined below

   Females do not need to use birth control during or following study drug treatment if considered of non-childbearing potential due to meeting any of the following criteria:
   * Postmenopausal, age ≤ 55 years with no menses for 12 or more months without an alternative medical cause AND an follicle stimulating hormone (FSH) level > 40 IU/L.
   * Permanently surgically sterile (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
5. Female who is not pregnant, breastfeeding, or considering becoming pregnant during the study or for approximately 120 days after the last dose of study drug.
6. Male subjects who are sexually active with a female partner of childbearing potential, must agree to use condoms, even if the male subject has undergone a successful vasectomy, from Study Day 1 through 120 days after the last dose of study drug. His female partner(s) must also use at least one of the following methods of birth control:

   * Combined (oestrogen and progestogen containing) hormonal birth control (oral, intravaginal, injectable, transdermal) associated with inhibition of ovulation initiated at least 30 days prior to study Baseline Day 1.
   * Progestogen-only hormonal birth control (oral, injectable, implantable) associated with inhibition of ovulation initiated at least 30 days prior to study Baseline Day 1.
   * Bilateral tubal occlusion/ligation.
   * Intrauterine device (IUD).
   * Intrauterine hormone-releasing system (IUS).
7. Male who is not considering fathering a child or donating sperm during the study or for approximately 120 days after the last dose of study drug.
8. Laboratory values meet the following criteria:

   * Serum aspartate transaminase (AST) and alanine transaminase (ALT) ≤ the upper limit of normal (ULN) at the Screening Visit and upon initial confinement.
   * Negative test result for hepatitis A virus immunoglobulin M (HAV-IgM), hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody (Ab) and human immunodeficiency virus (HIV) at screening visit.
   * Negative screen for drugs of abuse, alcohol or cotinine at screening and upon initial confinement.
   * For non-postmenopausal female subjects, a negative urine pregnancy test at the screening visit and a negative serum pregnancy test upon initial confinement and prior to the first dose of study drug.
   * No other laboratory results that the investigator determines are clinically significant.
   * Platelets greater than or equal to the lower limit of normal.
9. No clinically significant ECG abnormalities including

   * No evidence of 2nd or 3rd degree AV block at screening visit and upon initial confinement.
   * QT interval corrected for heart rate (QTc) using Fridericia's correction formula (QTcF) is ≤ 430 msec (males) or ≤ 450 msec (females) at screening visit and upon initial confinement.
10. A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG.
11. No history of: epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
12. No history of any clinically significant sensitivity or allergy to any medication or food.
13. No history of or active medical condition(s) or surgical procedure(s) that might affect gastrointestinal motility, pH, or absorption [e.g., Crohn's disease, celiac disease, gastroparesis, short bowel syndrome, gastric surgery (except pyloromyotomy for pyloric stenosis during infancy), cholecystectomy, vagotomy, bowel resection].
14. No evidence of dysplasia or history of malignancy (including lymphoma and leukemia) other than successfully treated non-metastatic cutaneous squamous cell, basal cell carcinoma or localized carcinoma in situ of the cervix.
15. No history of any clinically significant illness/infection/major febrile illness, hospitalization, or any surgical procedure within 30 days prior to the first dose of study drug.
16. Has not donated blood (including plasmapheresis), lost ≥ 550 mL blood volume, or received a transfusion of any blood product within 8 weeks prior to study drug administration.
17. No consumption of alcohol, grapefruit products, Seville oranges, starfruit products or quinine/tonic water within the 72-hour period prior to study drug administration.
18. No use of tobacco or nicotine-containing products within 180 days prior to the first dose of study drug.
19. No history of clinically significant (per Investigator's judgment) drug or alcohol abuse within the last 6 months.
20. Is not currently enrolled in another interventional clinical study.
21. Has not been previously enrolled in this study.
22. In the opinion of the investigator, this subject is a suitable candidate for enrollment in the study.
23. Subjects must not have been treated with any investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug.
24. Subject must not have received any live vaccine within 4 weeks prior to the first dose of study drug, or expected need of live vaccination during study participation including at least 4 weeks after the last dose of study drug.
25. Subject must not require any over-the-counter and/or prescription medication, vitamins and/or herbal supplements, with the exception of contraceptives or hormonal replacement therapies for females, on a regular basis.
26. Subject must not use any medications within the 2-week period prior to study drug administration.
27. Receipt of any drug by injection within 30 days or within a period defined by 5 half-lives, whichever is longer, prior to study drug administration.
28. No use of known inhibitors (e.g., ketoconazole) or inducers (e.g., carbamazepine) of cytochrome P450 3A (CYP3A) within 1 month prior to study drug administration.
29. No exposure to DSM265 within the past 90 days prior to first dose of study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Moehrle, Ass Prof, Study Director — Medicines for Malaria Venture; David Carter, MD, Principal Investigator — AbbVie Clinical Pharmacology Research Unit (ACPRU)
Locations (1):
- AbbVie Clinical Pharmacology Research Unit (ACPRU), Grayslake, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical Pharmacology phase 1 unit.
Pre-assignment Details: 30 day screening period.
Period: Overall Study
Arm/Group | DSM265 25% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fed
Started | 14 | 14 | 14
Completed | 14 | 14 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DSM265 25% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fed | Total
Number analyzed (Participants) | 14 | 14 | 14 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (10.78) | 36.1 (9.23) | 38.6 (10.58) | 37.6 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 9
  Male | 11 | 11 | 11 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 13 | 14 | 12 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 8 | 3 | 17
  White | 7 | 4 | 11 | 22
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 14 | 42

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Maximum observed DSM265 plasma concentration
Time Frame: 21 days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: NG/ML
Arm/Group | DSM265 25% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fed
Number analyzed (Participants) | 14 | 14 | 14
NG/ML | 15300 (27) | 14200 (28) | 11200 (27)
Statistical Analysis 1: Comparison: DSM265 25% SDD, 400 mg Fasted vs DSM265-TPGS 34% SDD, 400 mg Fasted; Test type: Equivalence — 2 comparisons performed: Reg. B vs. Reg. A, & Reg.C vs. Reg. B. Bioavailability of each test reg. relative to that of each reference reg. assessed via 90% CI. CI obtained by taking the antilog of the upper and lower limits of CI for the difference of the least squares means on the log scale within the ANOVA framework model. Bioequivalence between a test reg. and the reference reg. is concluded if the 90% CI from the analyses of the natural log of Cmax and AUC are within 0.80 to 1.25 range; p = 0.4847, ANOVA; Least Squares Means Log scale = 0.926, 90% CI 2-sided [0.771 to 1.113]
Statistical Analysis 2: Comparison: DSM265-TPGS 34% SDD, 400 mg Fasted vs DSM265-TPGS 34% SDD, 400 mg Fed; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0370, ANOVA; Least Squares Means Log scale = 0.790, 90% CI 2-sided [0.658 to 0.950]

2. Primary Outcome: AUC168
Description: Area under the plasma concentration-time curve from time 0 to 168 hours (AUC168)
Time Frame: 168 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: NG*H/ML
Arm/Group | DSM265 25% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fed
Number analyzed (Participants) | 14 | 14 | 14
NG*H/ML | 1100000 (14) | 987000 (17) | 1160000 (22)
Statistical Analysis 1: Comparison: DSM265 25% SDD, 400 mg Fasted vs DSM265-TPGS 34% SDD, 400 mg Fasted; Test type: Equivalence — Bioavailability of each test reg. relative to each reference reg will be assessed via 90% CI obtained from the analyses of the natural logs of Cmax and AUC. These CI are obtained by taking the antilog of the upper & lower CI for the difference of the least squares means on the log scale within the ANOVA model. Bioequivalence between a test reg and the respective reference reg will be concluded if the 90% CI from the analyses of the natural log of Cmax and AUC are within the 0.80 to 1.25 range; p = 0.1135, ANOVA; Sum of squares = 0.899, 90% CI 2-sided [0.805 to 1.004]
Statistical Analysis 2: Comparison: DSM265-TPGS 34% SDD, 400 mg Fasted vs DSM265-TPGS 34% SDD, 400 mg Fed; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.0192, ANOVA; Sum of squares = 1.175, 90% CI 2-sided [1.051 to 1.312]

3. Primary Outcome: AUCt
Description: AUC from time 0 until the last measurable concentration (AUCt),
Time Frame: 21 days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: NG*H/ML
Arm/Group | DSM265 25% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fed
Number analyzed (Participants) | 14 | 14 | 14
NG*H/ML | 1750000 (20) | 1570000 (19) | 1840000 (20)
Statistical Analysis 1: Comparison: DSM265 25% SDD, 400 mg Fasted vs DSM265-TPGS 34% SDD, 400 mg Fasted; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.1759, ANOVA; Sum of squares = 0.898, 90% CI 2-sided [0.787 to 1.024] — Regimen B to A
Statistical Analysis 2: Comparison: DSM265-TPGS 34% SDD, 400 mg Fasted vs DSM265-TPGS 34% SDD, 400 mg Fed; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.0496, ANOVA; Sum of squares = 1.172, 90% CI 2-sided [1.027 to 1.338] — Regimen C to B

4. Primary Outcome: Tmax
Description: Time to Cmax.
Time Frame: 21 days
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | DSM265 25% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fed
Number analyzed (Participants) | 14 | 14 | 14
Hours | 2.4 (1.4) | 2.1 (0.9) | 11.4 (8.4)
Statistical Analysis 1: Comparison: DSM265 25% SDD, 400 mg Fasted vs DSM265-TPGS 34% SDD, 400 mg Fasted; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Least Squares Means = -0.2857, 90% CI 2-sided [-3.4313 to 2.8599], Standard Error of Mean 1.866979
Statistical Analysis 2: Comparison: DSM265-TPGS 34% SDD, 400 mg Fasted vs DSM265-TPGS 34% SDD, 400 mg Fed; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Least Squares Means = 9.3571, 90% CI 2-sided [6.2115 to 12.5028], Standard Error of Mean 1.866979 — Regimen C to B

5. Primary Outcome: β
Description: Apparent terminal phase elimination rate constant
Time Frame: 21 days
Measure: Mean (Standard Deviation); unit: 1/H
Arm/Group | DSM265 25% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fed
Number analyzed (Participants) | 14 | 14 | 14
1/H | 0.00556 (0.00189) | 0.00531 (0.00154) | 0.00595 (0.00231)

6. Primary Outcome: C168
Description: Plasma concentration at 168 hours
Time Frame: 7 days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: NG/ML
Arm/Group | DSM265 25% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fed
Number analyzed (Participants) | 14 | 14 | 14
NG/ML | 4090 (25) | 3540 (25) | 4200 (24)
Statistical Analysis 1: Comparison: DSM265 25% SDD, 400 mg Fasted vs DSM265-TPGS 34% SDD, 400 mg Fasted; (ANOVA) will be performed for Tmax, the terminal phase elimination rate constant β, and the natural logarithms of Cmax, AUCt, AUC168, AUCinf, and C168. The model will include the effects for regimen. For the tests on regimen effects, the denominator sum of squares will be the residual sum of squares for error. Within the ANOVA modeling framework, the test regimen will be compared to the respective reference regimen by a test with a significance level of 0.05; Test type: Equivalence — Bioequivalence between a test regimen and the respective reference regimen will be concluded if the 90% confidence intervals from the analyses of the natural logarithms of Cmax and AUC are within the 0.80 to 1.25 range; p = 0.1745, ANOVA; Sum of squares = 0.866, 90% CI 2-sided [0.727 to 1.032]
Statistical Analysis 2: Comparison: DSM265-TPGS 34% SDD, 400 mg Fasted vs DSM265-TPGS 34% SDD, 400 mg Fed; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.1105, ANOVA — For tests on regimen effects, the denominator sum of squares is the residual sum of squares for error. Within the ANOVA modeling framework, the test regimen is compared to the respective reference regimen by a test with a significance level of 0.05; Sum of squares = 1.185, 90% CI 2-sided [0.995 to 1.411]

7. Secondary Outcome: AUCinf
Description: AUC from time 0 to infinity (AUCinf)
Time Frame: 21 days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: NG*H/ML
Arm/Group | DSM265 25% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fed
Number analyzed (Participants) | 14 | 14 | 14
NG*H/ML | 1960000 (29) | 1760000 (26) | 2040000 (23)
Statistical Analysis 1: Comparison: DSM265 25% SDD, 400 mg Fasted vs DSM265-TPGS 34% SDD, 400 mg Fasted; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.3100, ANOVA; LEAST SQUARES MEANS FOR LOGARITHMS. = 0.901, 90% CI 2-sided [0.759 to 1.069]
Statistical Analysis 2: Comparison: DSM265-TPGS 34% SDD, 400 mg Fasted vs DSM265-TPGS 34% SDD, 400 mg Fed; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.1619, ANOVA; LEAST SQUARES MEANS FOR LOGARITHMS. = 1.156, 90% CI 2-sided [0.974 to 1.371]

ADVERSE EVENTS:
Time Frame: All adverse events reported from the time of study drug administration until 30 days or 5 half-lives after discontinuation of study drug administration will be collected, whether solicited or spontaneously reported by the subject. In addition, serious adverse events and protocol-related non-serious adverse events will be collected from the time the subject signs the study-specific informed consent.
Arm/Group | DSM265 25% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fasted | DSM265-TPGS 34% SDD, 400 mg Fed
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT03637517/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT03637517/SAP_001.pdf